CLINICAL TRIAL: NCT06802627
Title: Influence of Prehabilitation on Postoperative Pulmonary Complications in Patient Undergoing Lung Resection Surgery
Brief Title: Prehabilitation for Lung Cancer Patients Undergoing Lung Resection
Acronym: Fit4LungNeo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Principal Investigator, Filipa Kendall, Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ethics Committee CHUSJ 52/2024
Record Dates: First submitted 2024-07-25; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer; Lung Resection
Keywords: Prehabilitation; Lung resection; Exercise training; Postoperative pulmonary complications; Respiratory muscle training; Education
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized at baseline into one of the four intervention - Control group (CG) receive an education session; inspiratory muscle training group (IMT-G) receive an education session plus inspiratory muscle training; expiratory muscle training group (EMT-G) receive an education session plus expiratory muscle training; global exercise training group (GET-G) receive an education session plus physical exercise training.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (CG) (Active Comparator): Control group will receive a single in-person preoperative education session at the Faculty of Sport of University of Porto, one week after the patient's inclusion in the study. The education session will be delivered for the patient and his/her caregiver or family member.
  The information that will be delivery is going to be focused on:
  * Lifestyle changes regarding nutrition and daily physical activity.
  * Abstinence of the additive behaviors smoking, alcohol, and drug consumption.
  * Personal hygiene care and hospital routines.
  * Importance of postoperative physiotherapy. A booklet summarizing the information provided at the education session will be delivered for all participants.
  Interventions: Other: Education session
- Inspiratory Muscle Training Group (IMT-G) (Experimental): The IMT-G will be submitted to an education session (equal to the CG) plus 2-weeks of inspiratory muscle training (IMT).
  After the education session, patients will start the IMT program that will last two weeks. The IMT will be 5 days/ week, lasting ~20 minutes, using the PowerBreath KH2 device. All sessions will start with 5 min of stretching exercises and then the IMT. In the first week, the intensity of the PowerBreath KH2 will be set at 50% of the maximal inspiratory pressure (with 12 breaths per minute), and it will be increasing by 10% in the second week (with 15 breaths per minute). Patients will be continuously monitored by an oximeter and modified Borg scale All IMT session will take place at São João Hospital.
  Interventions: Other: Education session; Other: Inspiratory muscle training group
- Expiratory Muscle Training Group (EMT-G) (Experimental): The EMT-G will be submitted to an education session (equal to the CG) plus 2-weeks of expiratory muscle training (EMT).
  After the education session, patients will start the EMT that will last two weeks, 5 days a week.
  The sessions will last ~20 minutes and will be structured as follows:
  * 5 minutes of stretching exercises
  * 8 minutes of abdominal resistance exercises (1st week: 2 exercises, 4 sets of 8 repetitions; 2nd week: 2 exercises, 4 sets of 10 repetitions)
  * 8 minutes of specific EMT using the Philips Respironics Threshold PEP device (Load: 20 cmH2O; 10 expirations for minute) Patients will be continuously monitored by an oximeter and modified Borg scale. All EMT session will take place at São João Hospital.
  Interventions: Other: Education session; Other: Expiratory muscle training group
- Global Exercise Training Group (GET-G) (Experimental): The GET-G will be submitted to an education session (equal to the CG) plus 2-weeks of physical exercise, 3 sessions per week, 45-60 minutes.
  The structure is:
  Warm-up 5 minutes of whole-body stretching exercises
  Main workout:
  -Aerobic: Week 1: 20 min of treadmill walking at 70% of the mean speed achieved on the 6-minute walk test and limited by 80% of the max theoretical heart rate. Week 2: 20 min of treadmill walking at 80% of the mean speed achieved on the 6-minute walk test and limited by 80% of the max theoretical heart rate.
  -Resistance Week 1: 8 exercises, 2 sets of 8-10 repetitions, using body weight and elastic bands. Week 2: 8 exercises, 2 sets of 10-12 repetitions, using body weight and elastic bands Coll-down: 5 min of whole-body stretching exercises, holding the point of feeling lightness discomfort for 15 seconds.
  Patients will be continuously monitored by an oximeter and modified Borg scale.
  Interventions: Other: Education session; Other: Global exercise training group

INTERVENTIONS:
Other: Education session — The information that will be delivery is going to be focused on:
  * Lifestyle changes regarding nutrition and daily physical activity.
  * Abstinence of the additive behaviors smoking, alcohol, and drug consumption.
  * Personal hygiene care and hospital routines.
  * Importance of postoperative physiotherapy. A booklet summarizing the information provided at the education session will be delivered for all participants.
Other: Inspiratory muscle training group — Education Session (described in the control group) Inspiratory muscle training (IMT) After the education session, patients will start the IMT program that will last two weeks.
  The IMT will be 5 days/ week, lasting 20 minutes, using the PowerBreath KH2 device. In the first week, the intensity of the PowerBreath KH2 will be set at 50% of the maximal inspiratory pressure (with 12 breaths per minute), and it will be increasing by 10% in the second week (with 15 breaths per minute). Patients will be continuously monitored by an oximeter and modified Borg scale
  Arms: Inspiratory Muscle Training Group (IMT-G)
Other: Expiratory muscle training group — Education Session (described in the control group) Expiratory muscle training (EMT)
  After the education session, patients will start the EMT that will last two weeks, 5 days a week. The sessions will last 20 minutes and will be structured as follows:
  4 minutes of total body stretching exercises 8 minutes of abdominal resistance exercises:
  1. First week: 2 exercises, 4 sets of 8 repetitions
  2. Second week: 2 exercises, 4 sets of 10 repetitions 8 minutes of specific EMT using the Philips Respironics Threshold PEP device (Load: 20 cmH2O; 10 expirations for minute) Patients will be continuously monitored by an oximeter and modified Borg scale.
  Arms: Expiratory Muscle Training Group (EMT-G)
Other: Global exercise training group — The GET-G will be submitted to an education session (equal to the CG) plus 2-weeks of physical exercise, 3 sessions per week, 45-60 minutes.
  The structure is:
  Warm-up: 5 minutes of whole-body stretching exercises
  Main workout:
  -Aerobic: Week 1: 20 min of treadmill walking at 70% of the mean speed achieved on the 6-minute walk test and limited by 80% of the max theoretical heart rate. Week 2: 20 min of treadmill walking at 80% of the mean speed achieved on the 6-minute walk test and limited by 80% of the max theoretical heart rate.
  -Resistance Week 1: 8 exercises, 2 sets of 8-10 repetitions, using body weight and elastic bands. Week 2: 8 exercises, 2 sets of 10-12 repetitions, using body weight and elastic bands Coll-down: 5 min of whole-body stretching exercises, holding the point of feeling lightness discomfort for 15 seconds.
  Patients will be continuously monitored by an oximeter and modified Borg scale.
  Arms: Global Exercise Training Group (GET-G)

SUMMARY:
Lung surgical resection is the gold standard treatment for earlier stages of lung cancer patients. Nevertheless, postoperative pulmonary complications (PPC) are frequent, related to morbidity and mortality, increasing length of hospital stay (LOS), hospital costs, delaying adjuvant treatments, and patients suffering. The PPC often occurs on postoperative days, even after hospital discharge. Prehabilitation might reduce PPC, although few studies have compared the effectiveness of different training protocols, and no information is available regarding the possible benefits of expiratory muscle training. Moreover, there are no comparisons of the cost-benefits of other protocols in patients submitted to lung resection surgery.

This project investigates the effectiveness of and compares four different prehabilitation protocols in reducing PPC and LOS in patients selected for lung cancer resections.

Participants will be individuals referred to surgical resection due to lung cancer. Patients who meet the inclusion criteria will be invited to participate in the study. After clinical data collection, patients will be randomly allocated (simple method) into four groups [Control - CG, receiving an education session; Inspiratory muscle training group (IMT-G) receiving education session plus inspiratory muscle training (IMT); expiratory muscle training group (EMT-G) receiving education session plus expiratory muscle training (EMT); global exercise training group (GET-G) receiving education session plus a general exercise training (GET)], and evaluated for functional capacity (pulmonary function, respiratory muscle function, physical fitness, daily physical activity, dyspnoea, fatigue, quality of life, anxiety, depression, and a 24-hour food diary. Afterward, all patients will receive an education class and written information regarding healthy habits to follow before, during, and after hospital discharge. Patients allocated to exercise groups will start the prehabilitation intervention for two weeks. After the intervention, patient assessments will be repeated. After that, patients will be submitted to surgery, and anesthetic and surgical procedure data will be collected. During hospital recovery, all patients will receive physiotherapy and any etiological complications and the LOS will be recorded according to medical criteria. After hospital discharge, PPC will be monitored and recorded for 30 days; by then, patients will be submitted to the final assessment.

DETAILED DESCRIPTION:
To achieve the project's aim, sample size was calculated using G*Power 3.1.9.2, based on an effect size of 0.33 reported by Cavalheri & Granger (2017) in a study of preoperative exercise training and pulmonary complications after lung resection. With α = 0.05 and 95% power, a sample of 180 patients (45 per group) was determined. Accounting for a 10% dropout rate, the estimated total sample size is 200 patients.

The study was approved by the Ethical Committee from the Unidade Local de Saúde de São João (ULS São João), number (52/2024). All patients who meet the inclusion criteria, selected for pulmonary resections due to lung cancer, will be invited to participate in the study at the first preoperative appointment at the Cardiothoracic Department of the ULS São João. After signing the informed consent statement, a cod number will be attributed to the patients to protect his/her personal information. Participants will be randomized into one of the four groups: control group (CG), inspiratory muscle training group (IMT-G), expiratory muscle training group (EMT-G), and global exercise group (GET-G).

Assessments will be conducted at three time points: after obtaining written informed consent (baseline), after completing the prehabilitation program (post-intervention), and 30 days post-discharge (follow-up). Each assessment will take two days.

First day of assessments (data collection at the hospital):

A physician will carry one a medical assessment and collect data regarding anthropometric, sociodemographic, medical history, and behavioral risk factors. Following the medical assessment, a researcher will provide to the patients an accelerometer to measure daily physical activity. The accelerometers will be worn during waking hours until completing the prehabilitation program. Additionally, the researcher will collect data regarding patient-related outcome measures through questionaries (modified Medical Research Council Dyspnoea Questionnaire, International Physical Activity Questionnaire - Short Form, the Fatigue Assessment Scale, the Hospital Anxiety and Depression Scale, the EuroQol 5D-5L, food intake report from the day before (1-day recall)]. Only in the baseline assessment, it will be placing the evaluation of barriers for prehabilitation. The researcher will then schedule the second day of assessment within the next three or four days.

Second day (data collection at Faculty of Sport of the University of Porto):

In the second day, patients will be evaluated for pulmonary function, respiratory muscle function, and functional capacity and physical fitness. Pulmonary function and respiratory muscle function will provide information on respiratory dynamics, including the absolute and predicted values of forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), peak expiratory flow (PEF), Tiffeneau index (TI); total lung capacity (TLC), diffusion lung capacity for carbon monoxide (DLCO) and DLCO per unit alveolar volume (DLCO/VA). Regarding respiratory muscle function, maximal voluntary ventilation (MVV), maximal inspiratory pressure (MIP), and maximal expiratory pressure (MEP) will be measured. Thereafter, patients will be assessed for functional capacity / physical fitness [aerobic endurance (6-minute walk test); lower body strength (30-second sit to stand), agility, coordination and dynamic balance (time up and go), balance (3 balance positions), speed walk (4 meters), lower body power (5-time sit to stand), handgrip strength].

One week after the acceptance in participating in the study, the intervention program will start with an in-person education session for all patients, and those from the IMT-G, EMT-G and GET-G will thereafter start their 2-week training interventions at ULS São João. Detailed information of the training interventions is described in the Arms and Interventions section.

Following the intervention, all patients will be reassessed using the same procedures as at baseline, and then they will undergo the surgery. Information on ASA classification, ARISCAT score, minimum oxygen saturation, surgical approach, total surgical time, and extent of resection will be registered by the surgical team.

After surgery, all patients will receive standard care at the Cardiothoracic Department, including daily medical assessment, physiotherapy care, and analgesic protocol. Postoperative pulmonary complications (PPC) or from any other etiology, as well as the length of hospital stay (LOS), will be recorded. Any postoperative complication and hospital readmission in the next 30 days will be monitored and recorded. The criteria of PPC will be established according to the European Society of Thoracic Surgery and the Society of Thoracic Surgeons joint agreement and standardized definition (Fernandez et al., 2015).

Following hospital discharge, patients will be referred for outpatient physiotherapy and nursing care. Three weeks post-discharge, patients will have a medical appointment at the Cardiothoracic Department and scheduled for the post-discharge assessment. At this appointment, patients will receive an accelerometer to wear for one week, after which a follow-up assessment will be conducted. At the end of data collection, a cost effective analysis will be perfumed aiming to achieve the real economic cost-benefit of each protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients accepted for lung resection surgery, due to lung cancer, at the Cardiothoracic Department of Unidade Local de Saúde São João
* Not included in any type of prehabilitation program

Exclusion Criteria:

* Diagnosis of cardiac, or hematological or neurologic diseases
* Pulmonary hypertension
* Renal failure
* Patients that underwent previous thoracic surgery
* Patients submitted to pneumectomy
* Patients with cognitive and mental disorders
* Patients with impairments in autonomous deambulation
* Patients already included in any prehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of postoperative pulmonary complications from surgery to 30 days after discharge | From the surgical procedure until 30 days after hospital discharge
  PPC according to the European Society of Thoracic Surgery and the Society of Thoracic Surgeons (Fernandez et al., 2015):
  * Persistent air leak > 5 days (thoracic drainage system Thopaz+ Medela)
  * Atelectasis needing bronchoscopy
  * Pneumonia
  * Adult respiratory distress syndrome
  * Bronchopleural fistula confirmed by CT scan or bronchoscopy
  * Pulmonary embolism confirmed by CT scan
  * Initial ventilator support > 48 hours
  * Reintubation
  * Tracheostomy
  * Empyema confirmed by CT scan
  * Chylothorax confirmed by CT scan and pleural liquid analysis
Length of hospital stay | From the surgical procedure until 30 days after hospital discharge
  The number of days of postoperative hospitalization including hospital readmissions related to surgery, assessed in clinical data. This will be based on the patients´ clinical files.

SECONDARY OUTCOMES:
Changes in pulmonary function from baseline at the day before surgery and for 1 week 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Absolute and relative values of Forced vital capacity (L) and (%); Forced Expiratory Volume in 1 second (L) and (%); Peak Expiratory Flow (L/s) and (%); Tiffeneau Index (%); Total Lung Capacity (L) and (%); Diffusion Lung Capacity for Carbon Monoxide (mmol/min/kPa) and (%); Diffusion Lung Capacity for Carbon Monoxide per unit alveolar volume (mmol/min/kPa/L) and (%) (MILLER et al., 2005). These informations will be captured using the equipment Quark PFT®, Cosmed (Rome, Italy)
Changes in respiratory muscle function from baseline at the day before surgery and for 1 week 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Absolute and relative values of Maximal Voluntary Ventilation (L/min) and (%); Maximal Inspiratory Pressure (cmH2O) and (%); Maximal Expiratory Pressure (cmH2O) and (%) ("ATS/ERS Statement on respiratory muscle testing," 2002).
  These informations will be captured using the equipment Quark PFT®, Cosmed (Rome, Italy)
  Baseline, day before surgery and 30 days after hospital discharge
Changes in aerobic endurance from baseline, at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Aerobic endurance will be assessed by the six-minute walk test (6-MWT), according to the American Thoracic Society (ATS) guidelines ("ATS statement: guidelines for the six-minute walk test," 2002). Distance (in meters), maximum and minimum oxygen saturation (%) and maximum and minimum heart rate (bpm) will be recorded. Both oxygen saturation and heart rates will be collected using the Spirodoc® (Rome, Italy).
Changes in lower body strength from baseline, at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  To measure lower body strength, participants will be required to perform the sit-to-stand test of the Senior Fitness Test (JONES, RIKLI & BEAM, 1999). Patients will be instructed to sit and stand the maximum times for 30 seconds. The total number of repetitions will be recorded.
Changes on handgrip strength from baseline, at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Handgrip strength will be assessed using the dynamometer Jamar Plus + Digital hand dynamometer (Sammons Preston Inc., Bolingbrook, Illinois, USA). Measurements will be carried out according to the American Society of Hand Therapists Recommendations (MacDermid et al., 2015). In brief, three measurements will be assessed in both arms, with 1 minute interval between attempts. The highest record for each arm will be used as the result.
Changes in balance from baseline, at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Balance will be measured by the balance test of the Short Physical Performance Battery. In brief, participants must stand for the maximum of 10 seconds with the two feet side by side, holding semitandem, or holding tandem (GURALNIK et al., 1994).
Changes in speed walk from baseline, at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge.
  Speed walk will be measured according to the Short Physical Performance Battery. To measure speed walk, participants must walk along 4 meters using their usual speed. Procedure will be performed 3 times (GURALNIK et al., 1994).
Changes in lower body power from baseline, at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge.
  Lower body power will be measured according to the Short Physical Performance Battery. Participants will be asked to stand up and sit down from an armless chair 5 times as fast as possible, and the time spend in the task will be record, and to (GURALNIK et al., 2000).
Changes in agility, coordination and dynamic balance from baseline, at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge.
  Agility, coordination and dynamic balance will be measured by the time up and go test presented in the Vivifrail battery (IZQUIERDO et al., 2016). The test will start with the participant sitting in a chair. At the evaluated sign, the participants will stand up, walk 3 meters, and turn back to the chair. The time to accomplish this task will be recorded.
Changes in dyspnea from baseline, at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  The modified Medical Research Council Dyspnea Questionnaire will be used to observed dyspnea. The questionary contains 5 sentences about daily activities that might promote dyspnea, and the participants will classify their self-perception of dyspnea according to a score ranging from 0 to 4 points (RIBEIRO et al., 2022).
Changes in fatigue from baseline, the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Fatigue will be determined through the Fatigue Assessment Scale, which is composed by 10 questions related to physical and mental fatigue, with a Lickert scale (1 to 5). The total score ranges from 10 to 50, which higher results indicating a more severe fatigue profile (MICHIELSEN et al., 2004).
Changes in anxiety and depression from baseline, the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Anxiety and depression will be evaluated with The Hospital Anxiety and Depression Scale. This scale consists of two subscales, one for anxiety and the other for depression. Higher results will indicate a potential presence of anxiety and depression (PAIS-RIBEIRO et al., 2007).
Changes in quality of life from baseline, the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Health-related quality of life will be observed with the EuroQol 5D-5L. This questionnaire contains the dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and participants also classified their perception of general health status (FENG et al., 2021).
Changes in objectively daily physical activity from baseline at the day before surgery and for 1 week 30 days after hospital discharge | From baseline to the day before surgery and for 1 week 30 days after hospital discharge
  Daily physical activity data will be objectively collected using GT3X+ accelerometers (ActiGraph®, LLC, Pensacola, FL, USA). The devices will be wearing for 8 hours during the waiting time for surgery and during 7 days after 30 days of hospital discharge. Data will be processed using the ActiLife software (ActiLife®, LLC, Pensacola, FL, USA).
Changes in subjective daily physical activity from baseline, at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  The Physical Activity Questionnaire - Short Form (IPAQ-SF) will be used to report subjective daily physical activity. Questions covering information about the weekly volume spent at vigorous, moderate and light physical activity, and the amount of time spending in the sitting position will be collected during the waiting time for surgery and during 7 days after 30 days of hospital discharge (CRAIG et al., 2003).
Change from Baseline on body composition at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Body composition variables (body mass (kg), fat-free mass (kg) and fat mass (kg)) will be analyzed with a bioimpedance (InBody 770®, InBody Co. Ltd., Seoul, South Korea).
Changes in body mass index from baseline at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Body mass index will be calculated by the formula: weight divided by squared height. Weight will be assessed with the scale InBody 770 ®, InBody Co. Ltd., Seoul, South Korea) and height with a wall mounted stadiometer.
Changes in food intake from baseline at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Registration of food intake, including alcohol consumption, will be determined with the 1-day food record. Data will be analyzed using the Food Processor Software®.
Changes in tabaco smoking habits from baseline at the day before surgery and 30 days after hospital discharge | Baseline, day before surgery and 30 days after hospital discharge
  Registration of smoking habits as "never smoker", "former smoker" or "smoker". For the "former smoker" and "smoker", it will be calculated the tabaco consumption by the number of pack year unity using the formula: number of cigarettes per day / 20 X number of smoking years (BERNAARDS et al., 2001).
Economic impact | Surgical procedure until 30 days after hospital discharge
  Specific costs attributed to each intervention and comparison cost-effectiveness of each program.

OTHER OUTCOMES:
Sociodemographic variables | Baseline
  Age (years), academic level (primary, secondary, bachelor, master, PhD), civil status (married, separated, widow, single, others). These will be assessed by interview.
Medical history | Baseline
  Diagnosed of diseases and number of medications will be assessed by one of the research members.
Barriers questionnaire for prehabilitation | Baseline
  Participation in a prehabilitation program might be difficult for the same patients due to many reasons, thus, to clarify barriers and in future develop solutions, all patients who fulfill inclusion criteria will be asked to answer the barriers questionnaire, even those who decline to participate in the clinical trial. The questionnaire has 21 questions with 5 possible answers and the last one in open version.

CONTACTS AND LOCATIONS:
Overall Officials: José F Oliveira, PhD, Study Chair — Faculty of Sport - University of Porto
Locations (1):
- Faculty of Sport - University of Porto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michielsen, H. J., De Vries, J., Van Heck, G. L., Van de Vijver, F. J. R., & Sijtsma, K. (2004). Examination of the Dimensionality of Fatigue: The Construction of the Fatigue Assessment Scale (FAS). European Journal of Psychological Assessment, 20(1), 39-48. https://doi.org/10.1027/1015-5759.20.1.39
- [Background] Izquierdo M, Casas-Herrero A, Zambom-Ferraresi F, Martínez-Velilla N, Alonso-Bouzón C, RodríguezMañas L. ViviFrail - A Practical Guide for Prescribing a Multi-Component Physical Training Program to prevent weakness and falls in People over 70. Multi-Component Physical Exercise Program Vivifrail, 2016. https://vivifrail.com/wp-content/uploads/2019/11/VIVIFRAIL-ENG-Interactivo.pdf
- [Background] Trost SG, McIver KL, Pate RR. Conducting accelerometer-based activity assessments in field-based research. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S531-43. doi: 10.1249/01.mss.0000185657.86065.98. PMID 16294116
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] Ribeiro S, Cardoso CS, Valerio M, Machado J, Costa J, Rodrigues C, Rebelo-Marques A. Confirmatory Evaluation of the Modified Medical Research Council Questionnaire for Assessment of Dyspnea in Patients with Chronic Obstructive Pulmonary Disease in Portugal. Acta Med Port. 2022 Feb 1;35(2):89-93. doi: 10.20344/amp.15208. Epub 2021 Apr 19. PMID 33877963
- [Background] Pais-Ribeiro J, Silva I, Ferreira T, Martins A, Meneses R, Baltar M. Validation study of a Portuguese version of the Hospital Anxiety and Depression Scale. Psychol Health Med. 2007 Mar;12(2):225-35; quiz 235-7. doi: 10.1080/13548500500524088. English, Portuguese. PMID 17365902
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] MacDermid J, Solomon G, Fedorczyk J, Valdes K. Clinical assessment recommendations 3rd edition: Impairment-based conditions. American Society of Hand Therapists; 2015. https://editions.mydigitalpublication.com/publication/?i=826932&p=2&view=issueViewer
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Fernandez FG, Falcoz PE, Kozower BD, Salati M, Wright CD, Brunelli A. The Society of Thoracic Surgeons and the European Society of Thoracic Surgeons general thoracic surgery databases: joint standardization of variable definitions and terminology. Ann Thorac Surg. 2015 Jan;99(1):368-76. doi: 10.1016/j.athoracsur.2014.05.104. PMID 25555970
- [Background] Feng YS, Kohlmann T, Janssen MF, Buchholz I. Psychometric properties of the EQ-5D-5L: a systematic review of the literature. Qual Life Res. 2021 Mar;30(3):647-673. doi: 10.1007/s11136-020-02688-y. Epub 2020 Dec 7. PMID 33284428
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Bernaards CM, Twisk JW, Snel J, Van Mechelen W, Kemper HC. Is calculating pack-years retrospectively a valid method to estimate life-time tobacco smoking? A comparison between prospectively calculated pack-years and retrospectively calculated pack-years. Addiction. 2001 Nov;96(11):1653-61. doi: 10.1046/j.1360-0443.2001.9611165311.x. PMID 11784461
- [Background] Cavalheri V, Granger C. Preoperative exercise training for patients with non-small cell lung cancer. Cochrane Database Syst Rev. 2017 Jun 7;6(6):CD012020. doi: 10.1002/14651858.CD012020.pub2. PMID 28589547
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180